CLINICAL TRIAL: NCT04927897
Title: DETECT: Defining the Target Volume for Endoluminal Radiation Boosting in Patients With Rectal Cancer
Brief Title: DETECT: Target Volume for Rectal Endoluminal Radiation Boosting
Acronym: DETECT
Status: Recruiting | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Maastricht University Medical Center (Other); Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Sponsor
Other Study IDs: NL77886.068.21
Record Dates: First submitted 2021-06-09; First posted 2021-06-16 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Rectal Cancer
Keywords: Rectal Cancer; Microscopic Tumor Spread; Target Volume Definition; Endoluminal Radiation Boosting
MeSH Terms: conditions — Rectal Neoplasms | interventions — Ultrasonography; Proctoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * The (re)biopsy material
  * (Part of) the material of the pathological rectal specimen after TME surgery
  Both are part of standard clinical care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: In addition to standard workup and treatment, patients will undergo pre-operatively, after induction of general anaesthesia, an endorectal ultrasound and rigid rectoscopy as study procedures if these are not part of standard workup yet.
  Interventions: Diagnostic Test: Ultrasound; Diagnostic Test: Rectoscopy; Other: Scan, e.g. CT (resection specimen)

INTERVENTIONS:
Diagnostic Test: Ultrasound — 3D endorectal ultrasound.
Diagnostic Test: Rectoscopy — Rigid rectoscopy.
Other: Scan, e.g. CT (resection specimen) — For some patients, images of the resection specimen (note: NOT of the patients) during the pathological process will be acquired.

SUMMARY:
The aim of the study is to provide prospective data regarding microscopic tumor spread in all directions from the macroscopic tumor in pathology specimens, as seen by eye, and on imaging to define the target volume for endoluminal radiation boosting in rectal cancer patients.

DETAILED DESCRIPTION:
This study is a prospective multicentre cohort trial in ≥50 patients with a residual ycT1-3N0 tumor after neoadjuvant chemoradiotherapy or radiotherapy for rectal adenocarcinoma at least 6 weeks after the neoadjuvant treatment.

In addition to standard workup and treatment (e.g. a flexible endoscopy and an MRI scan at 6-8 weeks post-neoadjuvant therapy), patients will undergo pre-operatively, after induction of general anaesthesia, an endorectal ultrasound and rigid rectoscopy as study procedures if these procedures are not already part of standard workup. Furthermore, the pathological specimens of some patients will be scanned using MR imaging during certain parts of the pathological process.

Objectives include determining the maximum distance of microscopic tumor spread per patient in all directions, creating a tissue deformation model to account for changes due to e.g. fixation and pathological processing, using this tissue deformation model to translate the microscopic tumor spread back to the in vivo situation (e.g. back to in vivo MRI scans, 3D endo-ultrasounds), and evaluating/determining risk factors for the presence and/or extent of microscopic tumor spread.

This data will be used for target volume definition in rectal endoluminal radiation boosting.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age and capable of giving informed consent.
* ycT1-3N0(*) residual(**) histology confirmed rectal adenocarcinoma after neoadjuvant radiotherapy or long-course chemoradiotherapy for which patients will undergo TME surgery.
* Minimal interval between end of neoadjuvant chemoradiotherapy or radiotherapy: 6 weeks.

(*)= as determined by clinical assessment (digital rectal examination, endoscopy with or without biopsy) and/or MRI. Biopsy/histology around the time of diagnosis is adequate; no biopsy/histology is needed after neoadjuvant therapy.

(**)= including tumor regrowths/local recurrence after an initial clinical complete response and a "watch and wait" approach. These patients will also be included after the local recurrence has been determined using endoscopy and/or MRI.

Exclusion Criteria:

* Patient has received brachytherapy as part of neoadjuvant treatment.
* <18 years of age or incapable of giving informed consent.
* Patient has not been treated with neoadjuvant radiotherapy or long-course chemoradiotherapy.
* Patient will not undergo TME surgery for a ycT1-3N0 residual histology confirmed rectal adenocarcinoma.
* Interval between end of neoadjuvant therapy and surgery is <6 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a limited (ycT1-3N0) residual tumor after neoadjuvant radiotherapy or long-course chemoradiotherapy for rectal adenocarcinoma.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-08-16 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Maximum distance of microscopic tumor spread per patient in all directions from the macroscopic tumor remnant in the pathology specimen | During post-resection pathological analysis (i.e. approximately 14 days post-resection)
  The maximum distance of microscopic tumor spread in all directions from the macroscopic remnant in the specimen will be measured per patient in millimeters by the pathology department in the pathologic resection specimens.

SECONDARY OUTCOMES:
Maximum distance of microscopic tumor spread per patient from the macroscopic tumor remnant in the pathology specimen, reported separately for MTS perpendicular to the bowel wall and for MTS parallel to the bowel wall | During post-resection pathological analysis (i.e. approximately 14 days post-resection)
  Measured per patient in millimeters by the pathology department in the pathologic resection specimens. Microscopic tumor spread perpendicular to the bowel wall and parallel to the bowel wall will be reported separately.
Maximum distance of microscopic tumor spread per patient in all directions from the macroscopic tumor remnant in the pathology specimen excluding ypT0 patients | During post-resection pathological analysis (i.e. approximately 14 days post-resection)
  Measured per patient in millimeters by the pathology department in the pathologic resection specimens. For this secondary outcome, this will be reported excluding all ypT0 patients.
Maximum distance of microscopic tumor spread per patient in all directions from the macroscopic tumor remnant in the pathology specimen only including patients with microscopic tumor spread | During post-resection pathological analysis (i.e. approximately 14 days post-resection)
  Measured per patient in millimeters by the pathology department in the pathologic resection specimens. For this secondary outcome, this will be reported only for patients with microscopic tumor spread.
Maximum distance of microscopic tumor spread per patient in all directions from the macroscopic tumor remnant in the pathology specimen only for patients with regrowths | During post-resection pathological analysis (i.e. approximately 14 days post-resection)
  Measured per patient in millimeters by the pathology department in the pathologic resection specimens. For this secondary outcome, this will be reported only for patients with regrowths.
Tissue deformation factor/model to compensate for tissue deformation due to removal of the specimen from the body, formalin fixation and tissue processing at the pathology department | The tissue deformation model will be created once all required data (e.g. MRI scans, rectoscopy images, endorectal ultrasound images) is available (approximately 14 days post-surgery for the final included patient).
  The deidentified images of the flexible endoscopy and in vivo MRI scan will be collected for the study. During the certain parts of the pathologic process, e.g. before and after fixation, MRIs of the pathological specimens of some of the patients will be made. These deidentified images of the specimens, together with e.g. the deidentified endoscopic, rectoscopic, ultrasound and in vivo MR images and possibly with optical images taken during pathological analysis, will be used to develop the deformation model.
  The flexible endoscopy and in vivo MRI scan are both taken approximately 6-8 weeks post-neoadjuvant treatment. The images of the rigid rectoscopy and 3D endorectal ultrasound are taken directly before TME surgery.
Maximum distance of microscopic tumor spread per patient in all directions from the macroscopic tumor remnant as seen by eye and/or on imaging | When the tissue deformation model is finished (approximately 3 months after all data for every patient is available). For the imaging time frames: please refer to the description.
  The tissue deformation factor/model and the location of the microscopic tumor spread in relation to the macroscopic remnant determined during pathological analysis, will be used to determine the maximum distance of microscopic tumor spread in relation to the macroscopic tumor as seen by eye (rectoscopically/endoscopically) and/or on imaging (endo-ultrasound, MRI) per patient in all directions.
  The flexible endoscopy and in vivo MRI scan are both taken approximately 6-8 weeks post-neoadjuvant treatment. The images of the rigid rectoscopy and 3D endorectal ultrasound are taken directly before TME surgery.
Treatment margin (in the various directions) relative to the macroscopic tumor to cover 90% and 95% of all microscopic tumor spread | Once the microscopic tumor spread is determined for all patients (approximately 14 days post-surgery for the final included patient), the treatment margins will be calculated.
  Distance that covers the microscopic tumor spread in all directions in millimeters for 90 and 95% of patients, including 95% confidence intervals, both reported including and excluding ypT0 patients. Reported both by eye and on imaging, for which among others the tissue deformation model will be used.
Evaluation of risk factors for the presence and/or the extent of microscopic tumor spread identified by the meta-analysis we performed | ypT stage is determined during post-resection pathological analysis (i.e. approximately 14 days post-resection). The time interval is determined at the day of surgery.
  These risk factors include pathological T stage after chemoradiation (ypT stage) and time interval between neoadjuvant chemoradiotherapy and surgery.

OTHER OUTCOMES:
Identification of potential risk factors for the presence and the extent of microscopic tumor spread not yet identified by our meta-analysis | Most are determined during post-resection path. analysis (approx. 14 days post-resection). ycT stage is determined approx. 6-10 weeks post-neoadjuvant treatment (multidisciplinary team), in vivo imaging is done approx 6-8 weeks post-neoadjuvant treatment
  Potential risk factors include among others ycT stage, regrowths/local recurrence, diameter, predominant histologic grade, tumor regression score/grade (pathologically), vascular invasion, lymphatic invasion, perineural invasion, microsatellite instability (MSI) and parameters related to in vivo MR imaging.
Analysis of (re)biopsy material | Biopsy material is obtained at time of diagnosis.
  This includes the biopsy material at time of diagnosis, and also the rebiopsy material for patients with tumor regrowths/local recurrence after an initial clinical complete response and a "watch and wait" approach. These (re)biopsies are a part of the standard diagnostic work-up. Part of this analysis will be performed during this study by reassessment of the histology of the biopsy material and/or if applicable the rebiopsy material.

CONTACTS AND LOCATIONS:
Overall Officials: Maaike Berbée, MD, PhD, Principal Investigator — Maastro; Evert Van Limbergen, MD, PhD, Principal Investigator — Maastro
Locations (3):
- Netherlands (3):
  - Maastro, Maastricht, Limburg
  - Maastricht University Medical Center, Maastricht, Limburg
  - Catharina Hospital, Eindhoven, North Brabant

IPD SHARING:
Plan to Share IPD: No
The data will not be shared with other researchers, however the following applies if patients have given specific, additional consent:
  If patients have consented to the use of leftover body material and/or data in further studies, the deidentified images (endoscopy, rectoscopy, ultrasound, in vivo MRIs and specimen MRIs) and pathological specimens/samples including (re)biopsies, and the accompanying data can be used for further scientific research related to rectal cancer by the investigators, including investigators from collaborating institutions, without requiring additional informed consent.

REFERENCES:
- [Background] van Gijn W, Marijnen CA, Nagtegaal ID, Kranenbarg EM, Putter H, Wiggers T, Rutten HJ, Pahlman L, Glimelius B, van de Velde CJ; Dutch Colorectal Cancer Group. Preoperative radiotherapy combined with total mesorectal excision for resectable rectal cancer: 12-year follow-up of the multicentre, randomised controlled TME trial. Lancet Oncol. 2011 Jun;12(6):575-82. doi: 10.1016/S1470-2045(11)70097-3. Epub 2011 May 17. PMID 21596621
- [Background] Sebag-Montefiore D, Stephens RJ, Steele R, Monson J, Grieve R, Khanna S, Quirke P, Couture J, de Metz C, Myint AS, Bessell E, Griffiths G, Thompson LC, Parmar M. Preoperative radiotherapy versus selective postoperative chemoradiotherapy in patients with rectal cancer (MRC CR07 and NCIC-CTG C016): a multicentre, randomised trial. Lancet. 2009 Mar 7;373(9666):811-20. doi: 10.1016/S0140-6736(09)60484-0. PMID 19269519
- [Background] Peeters KC, Marijnen CA, Nagtegaal ID, Kranenbarg EK, Putter H, Wiggers T, Rutten H, Pahlman L, Glimelius B, Leer JW, van de Velde CJ; Dutch Colorectal Cancer Group. The TME trial after a median follow-up of 6 years: increased local control but no survival benefit in irradiated patients with resectable rectal carcinoma. Ann Surg. 2007 Nov;246(5):693-701. doi: 10.1097/01.sla.0000257358.56863.ce. PMID 17968156
- [Background] Maas M, Beets-Tan RG, Lambregts DM, Lammering G, Nelemans PJ, Engelen SM, van Dam RM, Jansen RL, Sosef M, Leijtens JW, Hulsewe KW, Buijsen J, Beets GL. Wait-and-see policy for clinical complete responders after chemoradiation for rectal cancer. J Clin Oncol. 2011 Dec 10;29(35):4633-40. doi: 10.1200/JCO.2011.37.7176. Epub 2011 Nov 7. PMID 22067400
- [Background] Maas M, Nelemans PJ, Valentini V, Das P, Rodel C, Kuo LJ, Calvo FA, Garcia-Aguilar J, Glynne-Jones R, Haustermans K, Mohiuddin M, Pucciarelli S, Small W Jr, Suarez J, Theodoropoulos G, Biondo S, Beets-Tan RG, Beets GL. Long-term outcome in patients with a pathological complete response after chemoradiation for rectal cancer: a pooled analysis of individual patient data. Lancet Oncol. 2010 Sep;11(9):835-44. doi: 10.1016/S1470-2045(10)70172-8. Epub 2010 Aug 6. PMID 20692872
- [Background] Rijkmans EC, Cats A, Nout RA, van den Bongard DHJG, Ketelaars M, Buijsen J, Rozema T, Franssen JH, Velema LA, van Triest B, Marijnen CAM. Endorectal Brachytherapy Boost After External Beam Radiation Therapy in Elderly or Medically Inoperable Patients With Rectal Cancer: Primary Outcomes of the Phase 1 HERBERT Study. Int J Radiat Oncol Biol Phys. 2017 Jul 15;98(4):908-917. doi: 10.1016/j.ijrobp.2017.01.033. Epub 2017 Jan 20. PMID 28366579
- [Background] Sun Myint A, Smith FM, Gollins S, Wong H, Rao C, Whitmarsh K, Sripadam R, Rooney P, Hershman M, Pritchard DM. Dose Escalation Using Contact X-ray Brachytherapy After External Beam Radiotherapy as Nonsurgical Treatment Option for Rectal Cancer: Outcomes From a Single-Center Experience. Int J Radiat Oncol Biol Phys. 2018 Mar 1;100(3):565-573. doi: 10.1016/j.ijrobp.2017.10.022. Epub 2017 Oct 20. PMID 29229327
- [Background] Appelt AL, Ploen J, Harling H, Jensen FS, Jensen LH, Jorgensen JC, Lindebjerg J, Rafaelsen SR, Jakobsen A. High-dose chemoradiotherapy and watchful waiting for distal rectal cancer: a prospective observational study. Lancet Oncol. 2015 Aug;16(8):919-27. doi: 10.1016/S1470-2045(15)00120-5. Epub 2015 Jul 5. PMID 26156652
- [Background] Garant A, Magnan S, Devic S, Martin AG, Boutros M, Vasilevsky CA, Ferland S, Bujold A, DesGroseilliers S, Sebajang H, Richard C, Vuong T. Image Guided Adaptive Endorectal Brachytherapy in the Nonoperative Management of Patients With Rectal Cancer. Int J Radiat Oncol Biol Phys. 2019 Dec 1;105(5):1005-1011. doi: 10.1016/j.ijrobp.2019.08.042. Epub 2019 Aug 30. PMID 31476417
- [Background] Verrijssen AS, Opbroek T, Bellezzo M, Fonseca GP, Verhaegen F, Gerard JP, Sun Myint A, Van Limbergen EJ, Berbee M. A systematic review comparing radiation toxicity after various endorectal techniques. Brachytherapy. 2019 Jan-Feb;18(1):71-86.e5. doi: 10.1016/j.brachy.2018.10.001. Epub 2018 Nov 3. PMID 30396854
- [Background] Smith FM, Rao C, Oliva Perez R, Bujko K, Athanasiou T, Habr-Gama A, Faiz O. Avoiding radical surgery improves early survival in elderly patients with rectal cancer, demonstrating complete clinical response after neoadjuvant therapy: results of a decision-analytic model. Dis Colon Rectum. 2015 Feb;58(2):159-71. doi: 10.1097/DCR.0000000000000281. PMID 25585073
- [Background] Verrijssen AS, Guillem J, Perez R, Bujko K, Guedj N, Habr-Gama A, Houben R, Goudkade D, Melenhorst J, Buijsen J, Vanneste B, Grabsch HI, Bellezzo M, Paiva Fonseca G, Verhaegen F, Berbee M, Van Limbergen EJ. Microscopic intramural extension of rectal cancer after neoadjuvant chemoradiation: A meta-analysis based on individual patient data. Radiother Oncol. 2020 Mar;144:37-45. doi: 10.1016/j.radonc.2019.10.003. Epub 2019 Nov 9. PMID 31710942
- [Background] Maas M, Lambregts DM, Nelemans PJ, Heijnen LA, Martens MH, Leijtens JW, Sosef M, Hulsewe KW, Hoff C, Breukink SO, Stassen L, Beets-Tan RG, Beets GL. Assessment of Clinical Complete Response After Chemoradiation for Rectal Cancer with Digital Rectal Examination, Endoscopy, and MRI: Selection for Organ-Saving Treatment. Ann Surg Oncol. 2015 Nov;22(12):3873-80. doi: 10.1245/s10434-015-4687-9. Epub 2015 Jul 22. PMID 26198074
- [Background] Nuernberg D, Saftoiu A, Barreiros AP, Burmester E, Ivan ET, Clevert DA, Dietrich CF, Gilja OH, Lorentzen T, Maconi G, Mihmanli I, Nolsoe CP, Pfeffer F, Rafaelsen SR, Sparchez Z, Vilmann P, Waage JER. EFSUMB Recommendations for Gastrointestinal Ultrasound Part 3: Endorectal, Endoanal and Perineal Ultrasound. Ultrasound Int Open. 2019 Jan;5(1):E34-E51. doi: 10.1055/a-0825-6708. Epub 2019 Feb 5. PMID 30729231
- [Background] Martens MH, Maas M, Heijnen LA, Lambregts DM, Leijtens JW, Stassen LP, Breukink SO, Hoff C, Belgers EJ, Melenhorst J, Jansen R, Buijsen J, Hoofwijk TG, Beets-Tan RG, Beets GL. Long-term Outcome of an Organ Preservation Program After Neoadjuvant Treatment for Rectal Cancer. J Natl Cancer Inst. 2016 Aug 10;108(12):djw171. doi: 10.1093/jnci/djw171. Print 2016 Dec. PMID 27509881
- [Background] Simpson G, Hopley P, Wilson J, Day N, Haworth A, Montazeri A, Smith D, Titu L, Anderson J, Agbamu D, Walsh C. Long-term outcomes of real world 'watch and wait' data for rectal cancer after neoadjuvant chemoradiotherapy. Colorectal Dis. 2020 Nov;22(11):1568-1576. doi: 10.1111/codi.15177. Epub 2020 Jul 20. PMID 32686268
- [Background] Lam D, Kaneko Y, Scarlett A, D'Souza B, Norris R, Woods R. The Effect of Formalin Fixation on Resection Margins in Colorectal Cancer. Int J Surg Pathol. 2019 Oct;27(7):700-705. doi: 10.1177/1066896919854159. Epub 2019 Jun 14. PMID 31195869
- [Background] Kapali AS, Chandramohan K, Jayasudha AV. A Prospective Study of Distal Microscopic Spread in Rectal Cancer After Neoadjuvant Chemoradiation in Pinned and Unpinned Specimen. Indian J Surg Oncol. 2017 Dec;8(4):469-473. doi: 10.1007/s13193-017-0637-2. Epub 2017 Mar 18. PMID 29203975
- [Background] Park HS, Lee S, Haam S, Lee GD. Effect of formalin fixation and tumour size in small-sized non-small-cell lung cancer: a prospective, single-centre study. Histopathology. 2017 Sep;71(3):437-445. doi: 10.1111/his.13237. Epub 2017 Jun 16. PMID 28407385
- [Background] Goldstein NS, Soman A, Sacksner J. Disparate surgical margin lengths of colorectal resection specimens between in vivo and in vitro measurements. The effects of surgical resection and formalin fixation on organ shrinkage. Am J Clin Pathol. 1999 Mar;111(3):349-51. doi: 10.1093/ajcp/111.3.349. PMID 10078110
- [Background] Tran T, Sundaram CP, Bahler CD, Eble JN, Grignon DJ, Monn MF, Simper NB, Cheng L. Correcting the Shrinkage Effects of Formalin Fixation and Tissue Processing for Renal Tumors: toward Standardization of Pathological Reporting of Tumor Size. J Cancer. 2015 Jul 2;6(8):759-66. doi: 10.7150/jca.12094. eCollection 2015. PMID 26185538
- [Background] Dayde D, Tanaka I, Jain R, Tai MC, Taguchi A. Predictive and Prognostic Molecular Biomarkers for Response to Neoadjuvant Chemoradiation in Rectal Cancer. Int J Mol Sci. 2017 Mar 7;18(3):573. doi: 10.3390/ijms18030573. PMID 28272347
- [Background] Thies S, Langer R. Tumor regression grading of gastrointestinal carcinomas after neoadjuvant treatment. Front Oncol. 2013 Oct 7;3:262. doi: 10.3389/fonc.2013.00262. PMID 24109590